CLINICAL TRIAL: NCT06491888
Title: A Multicenter Randomized Controlled Study of Fluorescence Photoelectric Cervical Lesion Image Detector in Cervical Cancer Screening
Brief Title: A Multicenter Randomized Controlled Study of Photoelectric Detection in Cervical Cancer Screening
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Lei Li (Other)
Responsible Party: Sponsor-Investigator, Lei Li, Chief physician, Peking Union Medical College Hospital
Organization: Peking Union Medical College Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Screening
Other Study IDs: OITS2
Record Dates: First submitted 2024-07-01; First posted 2024-07-09 (Actual); Last update posted 2024-08-15 (Actual); Status verified 2024-08

CONDITIONS: Uterine Cervical Cancer; Cervical Intraepithelial Neoplasia; High Grade Squamous Intraepithelial Lesions; Low Grade Squamous Intraepithelial Lesions
MeSH Terms: conditions — Uterine Cervical Neoplasms; Uterine Cervical Dysplasia; Squamous Intraepithelial Lesions

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group Accepting Photoelectric Detection (Experimental): The subjects in this group need to undergo the detection of fluorescence photoelectric cervical lesion image detector before colposcopy, and then undergo routine colposcopy and biopsy after the detection.
  Interventions: Diagnostic Test: Detection of Cervical Lesions by Fluorescence Photoelectric Image
- Routine colposcopy group (No Intervention): Subjects who entered this group underwent colposcopy and biopsy according to the routine gynecological examination procedure.

INTERVENTIONS:
Diagnostic Test: Detection of Cervical Lesions by Fluorescence Photoelectric Image — Photoelectric detection was carried out on the subjects of the experimental group.
  Arms: Group Accepting Photoelectric Detection

SUMMARY:
The main purpose of this study is to verify the accuracy of the fluorescence photoelectric cervical lesion image detector relative to the pathological gold standard and the detection rate of CIN 2 +, as well as the significance of it as a shunt tool before colposcopy through a randomized controlled study.

The secondary objectives were to compare the relative pathological accuracy of the fluorescence photoelectric cervical lesion image detection results with the HPV detection results and cytological results, and to compare the lesion area displayed by the fluorescence photoelectric cervical lesion image detector with the lesion area that appeared after traditional colposcopy chemical staining.

In this study, 4200 subjects who have been evaluated and can be enrolled (these subjects have the indication of referral to colposcopy) will be included in the study, and they will be divided into two groups according to the principle of randomization. The histological results were obtained after routine colposcopy and biopsy. The experimental group first underwent colposcopy and biopsy after the judgment of the fluorescent photoelectric cervical lesion image detector to obtain histological results. Finally, the accuracy of the relative pathological results, the detection rate of CIN2 +, negative predictive value and positive predictive value of the two groups were compared.

ELIGIBILITY:
Inclusion Criteria:

* 1. Age ≥ 18 years old, ≤ 65 years old, with a complete cervix without deformity.
* 2. Have clear cervical cancer screening results, meet HPV16/18 (+) or high-risk HPV (+), and cervical cytology results ≥ ASC-US.
* 3. Fully informed and agreed to participate in the study.
* 4. No history of cervical cancer disease and cancer in other parts.

Exclusion Criteria:

* 1. Cannot meet all Inclusion Criteria.
* 2. There is clear immunosuppression, such as HIV infection or organ transplantation, etc., and the vagina or cervix is in the acute inflammation stage。
* 3. There are serious bleeding diseases or photosensitive diseases such as abnormal coagulation.

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4200 (Estimated)
Dates: Start 2024-08 (Estimated); Primary Completion 2025-07 (Estimated); Study Completion 2025-07 (Estimated)

PRIMARY OUTCOMES:
Sensitivity and specificity of a fluorescence photoelectric image detector for cervical lesions. | Enrolled subjects receive histopathological results approximately 7 days after colposcopy.
  Sensitivity and specificity of the fluorescence photoelectric detection technique relative to histopathological findings.
Detection rate of CIN2+ by fluorescence photoelectric cervical lesion image detector. | Enrolled subjects receive histopathological results approximately 7 days after colposcopy.
  The sensitivity, specificity, CIN2+ detection rate, negative predictive value and positive predictive value were compared between the fluorescence photoelectric technology and HPV detection results and cytology results, and the consistency and coincidence between the fluorescence photoelectric technology and HPV detection results and cytology results were calculated.

SECONDARY OUTCOMES:
The correlation between fluorescence photoelectric technology and HPV detection and cytology results. | Enrolled subjects receive histopathological results approximately 7 days after colposcopy.
  The sensitivity, specificity, CIN2+ detection rate, negative predictive value and positive predictive value were compared with the results of HPV detection and cytology.

CONTACTS AND LOCATIONS:
Locations (1):
- Lei Li, Beijing, Beijing Municipality, China